CLINICAL TRIAL: NCT06864312
Title: Mitigating Rebound Pain Following Regional Anaesthesia for Ankle Fracture Surgery: a Three-armed Randomised Control Trial
Brief Title: Rebound Pain Following Regional Anaesthesia for Ankle Fracture Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Brian Declan O'Donnell, Consultant Anaesthesiologist and Clinical Senior Lecturer, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANKLE 2023
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Ankle Fracture (bimalleolar Equivalent, Bimalleolar, or Trimalleolar); Ankle Fracture - Lateral Malleolus; Ankle Fracture - Medial Malleolus; Rebound Pain
Keywords: Rebound Pain; Ankle Fracture; Regional Anaesthesia; Nerve Block; Analgesia
MeSH Terms: conditions — Ankle Fractures; Agnosia | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Patients randomised to this group will receive the current 'gold standard' of post operative analgesic care: Popliteal Fossa Sciatic Block with standard postoperative multimodal analgesia
- Intervention Continuous Popliteal Fossa Sciatic Block (Experimental): Patients randomised to this group will receive standard of post operative analgesic care: Popliteal Fossa Sciatic Block with standard postoperative multimodal analgesia, together with a paraneural sciatic catheter placed at the time of block and used for the continuous postoperative administration of local anaesthetic
  Interventions: Drug: continuous infusion of levobupivacaine
- Intervention Timed opioid (Experimental): Patients randomised to this group will receive standard of post operative analgesic care: Popliteal Fossa Sciatic Block with standard postoperative multimodal analgesia, together with a timed (to coincide with expected nerve block offset) and weight appropriate dose of immediate release oxycodone.
  Interventions: Drug: oxycodone

INTERVENTIONS:
Drug: continuous infusion of levobupivacaine — patients one arm of this study will receive a postoperative continuous infusion of levobupivacaine
  Arms: Intervention Continuous Popliteal Fossa Sciatic Block
Drug: oxycodone — A timed weight appropriate dose of oxycodone will be administered 16 hours postoperatively
  Arms: Intervention Timed opioid

SUMMARY:
Regional anaesthesia is a commonly used and effective analgesic modality in orthopaedic surgery. The benefits of peripheral nerve blocks (PNB) include better pain relief, limited opioid consumption and high patient satisfaction(1-3).

Following ankle fracture surgery, rebound pain has been reported. The rebound effect was demonstrated in a randomised control trial comparing pain after ankle fracture repair under general anaesthesia with or without PNB(4). An increase in pain scores was demonstrated after PNB resolution exceeding that of the group without PNB. Prospective research from Cork University Hospital (CUH) in recent years has identified rebound pain as a clinically significant issue. 2018 CUH data have demonstrated that pain following ankle fracture surgery is well managed by PNB, with no reported pain until block regression(5). Upon block regression (12-18 hours postoperatively), the median pain score was 8 out of 10 on the numerical rating scale. Median peak pain score across all patients in the first 24 hours after block administration was 7.5.

Acute postoperative pain is an important problem due to negative patient consequences which include: increased morbidity; impaired physical function; prolonged hospital stay; and persistent pain. Studies to evaluate solutions to rebound pain are lacking. Favourable outcomes may be obtained with either continuous PNB(6) and timed systemic analgesics. Formal evaluation of such bespoke analgesic pathways is required.

We aim to establish an evidence-based strategy to prevent rebound pain. On a patient level, this would reduce the patient's experience of severe acute postoperative pain. This would improve a myriad of short- and long- term patient factors including; patient experience, opioid requirement, mobility, length of stay, chronic pain(7, 8). Rebound pain has additionally been reported following upper limb surgery(9). The knowledge generated by this study also has the potential to impact the postoperative analgesic management of upper limb fracture surgeries. This study aims to answer an original research question which has not been addressed in the literature to-date.

DETAILED DESCRIPTION:
Study objective To evaluate the effect of analgesic pathways on rebound pain following ankle fracture surgery. The hypothesis is that the intervention will reduce rebound pain by 50% on a numerical rating scale (0-10).

Methods

Trial design Three-armed randomised control trial.

Participants Inclusion criteria Patients undergoing surgery for ankle fracture ORIF receiving regional anaesthesia for postoperative analgesia.

Exclusion criteria Pain preoperatively of any source requiring analgesic consumption (on more than three occasions) within three months of surgery.

History of chronic pain syndrome. History of peripheral neuropathy. Clinically significant cognitive impairment (MiniMental state score < 24).

Interventions After giving written consent, patients will be assigned to one of 3 study groups using a random number generator.

All patients will receive standardised single shot ultrasound guided popliteal and sciatic nerve blocks.

Single shot peripheral nerve block standardised protocol 10ml of Bupivacaine 0.5% with 5ml of 2% lignocaine will be used in the popliteal sciatic block and 10ml of Bupivacaine 0.5% with 5ml of 2% lignocaine will be used in the saphenous block.

A lateral approach and subparaneural technique will be applied for the popliteal block at the level of the sciatic nerve bifurcation.

The saphenous block will be administered at the mid-femoral level. For patients who weigh less than 50kg, 10ml of Bupivacaine 0.25% with 5ml of 1% lignocaine will be used in the popliteal sciatic block and 10ml of Bupivacaine 0.25% with 5ml of 1% lignocaine will be used in the saphenous block.

General anaesthesia standardised protocol All patients will have standard monitoring applied intraoperatively. General anaesthesia will be administered using a regimen of intravenous fentanyl 1 mcg/kg, intravenous propofol 2-3 mg/kg and sevoflurane delivered in an oxygen / air mixture, or intravenous fentanyl 1 mcg/kg and total intravenous anaesthesia (TIVA) using a continuous propofol infusion Intravenous ondansetron 4mg, dexamethasone 8 mg, paracetamol 1g, and diclofenac 75 mg will be administered intraoperatively.

Postoperative analgesic plans will differ between groups as follows:

Group C: Postoperative oral analgesia as per current practice standardised protocol Regular paracetamol 1g six-hourly. Ibuprofen 400mg TDS, if not contraindicated. Oxycodone immediate release (Oxynorm) 10mg as required every 4 to 6 hours.

Group TO: timed opioid analgesia protocol Participants will receive single shot peripheral nerve block. Regular paracetamol QDS, regular ibuprofen 400mg TDS, if not contraindicated. Oxycodone immediate release (Oxynorm) 10mg as required every 4 to 6 hours. At 16 hours after block administration: "timed dose"of 10mg Oxynorm to be administered.

Group SC: Sciatic catheter protocol Following administration of the single shot nerve block, a peripheral catheter will be inserted under ultrasound guidance at the level of the sciatic bifurcation.

A continuous infusion of 0.25% bupivacaine at 5ml/hr will be commenced postoperatively on emergence of anaesthesia until 24 hours after PNB administration, at which time the catheter is to be removed.

A standard catheter-through-needle technique will be used for all patients and a regional-specific soft-tipped catheter left in situ with a filter attached. The continuous local anaesthetic will be infused via a standard mechanical wound infiltration pump. This is a 350ml hardshell pump which can provide consistent flow rates. It is non compressible and cannot cause excess dosage due to compression.

Regular paracetamol 1g six-hourly. Ibuprofen 400mg TDS, if not contraindicated. Oxycodone immediate release (Oxynorm) 10mg as required every 4 to 6 hours for breakthrough pain

Follow-up Patients will record changes in pain scores on diary sheets. Total PRN analgesia administered will be recorded from the bedside drug chart and patient pain diary.

QoR9 Questionnaire will be completed on ward or by telephone on Day 1 and Day 2 post-op.

On the same telephone call, participants will be asked to state peak pain score experienced in preceding 24 hours and will be asked to post back pain diaries.

Group SC will receive an information sheet about peripheral nerve block catheter care prior to discharge. The sheet will include contact details for the Regional Anaesthesia Fellow and Anaesthetics Senior Reg, should participants have any queries.

For Group SC, any catheter complications experienced will be recorded at 24 and 48 hours on ward/ by telephone.

Complications:

Catheter falling out <24 hours New swelling along the catheter track New tenderness around the catheter site New redness around the catheter site Block effects lasting more than 72 hours after removal of catheter New onset of weakness/ numbness 24 hours after the original block wears off If the entire catheter is not removed Outcomes

Primary outcome:

Median peak pain score in 24 hours after PNB administration.

Secondary outcomes:

Time of peak pain occurrence. Impact of intervention on quality of recovery. Defined population at highest risk of rebound pain.

Randomisation After giving written consent, patients will be assigned to one of 3 study groups using a random number generator.

Sample size Our data will be analysed using the ANOVA test to compare mean pain scores between groups. We will power our study to 95% and will set the significance level at 0.05. We hypothesise that our effect size will be 50%. This results in a required sample size of 22 patients in each arm. To allow for participants discontinuing enrolment and not responding to 24 and 48 hour follow-up we will enrol 37 patients in each arm of the study. Our total sample size will be 111.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for ankle fracture ORIF receiving regional anaesthesia for postoperative analgesia.

ASA Grades 1-3

Exclusion Criteria:

* Pain preoperatively of any source requiring analgesic consumption (on more than three occasions) within three months of surgery.

Open fractures Multiple injuries History of chronic pain syndrome. History of peripheral neuropathy. Clinically significant cognitive impairment (MiniMental state score < 24) Severe cardiac, respiratory, renal or endocrine dysfunction Allergy to any of the following: Lignocaine, Bupivacaine, Paracetamol, Diclofenac, Oxycodone, Dexamethasone, Propofol, Vecuronium.

Malignant Hyperthermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Rebound Pain | 17-24 hours following the ankle fracture surgery
  Patient reported pain on a 11 point (0-10) verbal rating pain scale upon regression of popliteal sciatic block or pain measured at a time point between 17-24 hours following the ankle fracture surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D O'Donnell, MBBChBAO MSc FCARCSI MD, Principal Investigator — Cork University Hospital & University College Cork
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided